CLINICAL TRIAL: NCT02586350
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Compare the Efficacy and Safety of Anlotinib Versus Placebo in Patients With Medullary Thyroid Carcinoma(ALTER01031)
Brief Title: Study of Anlotinib in Patients With Medullary Thyroid Carcinoma(ALTER01031)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-01-IIMTC
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Medullary Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent.Subjects with confirmation of disease progression by independent imaging review, while receiving blinded study drug may request to receive open label Anlotinib and enter the Optional Open Label Anlotinib Treatment Period of the Extension Phase. Subjects who request to receive open label Anlotinib(at the time of confirmed progression) will be informed whether they received placebo or Anlotinib during the period of blinded study drug administration. Subjects who received Anlotinib will not be eligible for the open-label phase.
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent.Subjects with confirmation of disease progression by independent imaging review, while receiving blinded study drug may request to receive open label Anlotinib and enter the Optional Open Label Anlotinib Treatment Period of the Extension Phase. Subjects who request to receive open label Anlotinib(at the time of confirmed progression) will be informed whether they received placebo or Anlotinib during the period of blinded study drug administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib
  Other Names: Anlotinib p.o. qd
  Arms: Anlotinib
Drug: Placebo — Placebo p.o. qd
  Arms: Placebo

SUMMARY:
To compare the effects and safety of Anlotinib with placebo in patients with Medullary Thyroid Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Histological documentation of medullary thyroid carcinoma(MTC),Unable to surgery(Stage IV) or metastasis ,With measurable disease (using RECIST1.1)
3. ECOG PS:0-1,Life expectancy of more than 6 months
4. main organs function is normal

Exclusion Criteria:

1. Prior treatment with Anlotinib or VEGFR-targeted therapies(such as Vandetanib,Cabozantinib,Lenvatinib,Sunitinib,Sorafenib etc.)
2. Subjects received radiotherapy external exposure within 3 months prior to the first dose of study drug or plan to be received any anti-cancer treatment during study
3. Patients suffering from other malignancies currently or within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancers and superficial bladder cancer [ Ta (non-invasive carcinoma), Tis (carcinoma in situ) and T1 (carcinoma invasion into lamina propria) ]
4. CTCAE(4.0) Grade 1 or higher non-remission toxicity induced by any other previous treatments，excluding alopecia and Grade 2 or lower neurotoxicity induced by oxaliplatin
5. Patients with factors that could affect oral medication (such as dysphagia etc.)
6. Patients with pleural effusion or ascites, causing respiratory syndrome (CTCAE Grade 2 or higher dyspnea [Grade 2 dyspnea refers to Shortness of breath with a small amount of activities, affecting Instrumental activities of daily life])
7. Patients underwent major surgical treatment，open biopsy or significant traumatic injury within 28 days prior to assignment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-07; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Date of randomization to the date of disease progression (measured every 6 weeks) or death (whichever occurs first) as determined by blinded independent imaging review(assessed up to 24 months)
  To compare the Progression-free Survival (PFS) of subjects with medullary thyroid carcinoma(MTC) with Anlotinib versus Placebo.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Date of randomization to the date of disease progression (measured every 6 weeks) or death (assessed up to 24 months)
  To compare Overall Response Rate (ORR) (Complete and Partial Responses, CR and PR) of subjects treated with Anlotinib versus Placebo.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guozhou, Guangdong
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - Henan Province Tumor Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - Jiangsu province tumor hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Of Sichuan University, Chongqing, Sichuan
  - 20th Floor, Block C, Lake Road, Hexi District, Tianjin Medical University Cancer Institute and Hospital ., Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang